CLINICAL TRIAL: NCT01366950
Title: Work Place Health Promotion as a Change Project
Brief Title: Work Place Health Promotion: a Change Project
Acronym: HEALTHCHANGE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Just Bendix Justesen, Ph.d. student, University of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: S-20110051
Record Dates: First submitted 2011-06-02; First posted 2011-06-06 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Health Prevention
MeSH Terms: interventions — Efficiency

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Excercise group (Experimental)
  Interventions: Behavioral: Intelligent physical activity
- Reference (No Intervention)

INTERVENTIONS:
Behavioral: Intelligent physical activity — 30 minutes of moderate activity 6 days a week and 45 minutes of high intensity training 1 day a week. Moderate activity is monitored in diaries and high intensity training is monitored by a trainer.
  Other Names: Change project; Productivity
  Arms: Excercise group

SUMMARY:
The purpose of this study is to determine if intelligent physical exercise training can increase the productivity of office workers in Denmark. Effects of intervention is measured after 1 and 2 years.

The project is driven as a change project.

The investigators measure productivity as:

* Individual health
* Sick leave
* Retention at the workplace

ELIGIBILITY:
Inclusion Criteria:

* Office workers

Exclusion Criteria:

* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2011-06; Primary Completion 2013-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
aerobic capacity | After 1 and 2 years

SECONDARY OUTCOMES:
sick leave | After 1 and 2 years
Individual productivity | After 1 and 2 years
Retention | After 1 and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Sjoegaard, Professor, Study Director — University of Southern Denmark
Locations (5):
- Denmark (5):
  - Nestlé, Copenhagen
  - Esbjerg Municipality, Esbjerg
  - National Board of Social Sciences, Odense and Copenhagen
  - TDC, Sønderborg
  - Varde Kommune, Varde

REFERENCES:
- [Derived] Christiansen HJ, Sogaard K, Justesen JB, Sjogaard G, Dalager T. Long Term Cardiovascular Health Effects of Intelligent Physical Exercise Training Among Office Workers-A 2 Year Follow up of a Randomized Controlled Trial. J Occup Environ Med. 2023 Oct 1;65(10):813-819. doi: 10.1097/JOM.0000000000002892. Epub 2023 May 23. PMID 37231634
- [Derived] Justesen JB, Sogaard K, Dalager T, Christensen JR, Sjogaard G. The Effect of Intelligent Physical Exercise Training on Sickness Presenteeism and Absenteeism Among Office Workers. J Occup Environ Med. 2017 Oct;59(10):942-948. doi: 10.1097/JOM.0000000000001101. PMID 28800039
- [Derived] Sjogaard G, Justesen JB, Murray M, Dalager T, Sogaard K. A conceptual model for worksite intelligent physical exercise training--IPET--intervention for decreasing life style health risk indicators among employees: a randomized controlled trial. BMC Public Health. 2014 Jun 26;14:652. doi: 10.1186/1471-2458-14-652. PMID 24964869